CLINICAL TRIAL: NCT03922308
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-blind Study in Patients With Acquired Thrombotic Thrombocytopenic Purpura (aTTP) to Evaluate the Pharmacokinetics, Safety and Efficacy of rADAMTS-13 (SHP655) Administered in Addition to Standard Of Care (SoC) Treatment
Brief Title: Study of rADAMTS-13 (SHP655) in the Treatment of Participants With Acquired Thrombotic Thrombocytopenic Purpura (aTTP)
Acronym: SOAR-HI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP655-201; 2018-003775-35 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2019-04-19 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura (aTTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of Care (SoC) + Placebo (Placebo Comparator): Participants received SoC daily PEX followed by placebo immediately and 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
  Interventions: Other: Placebo; Other: Standard of Care
- SoC + SHP655 + Placebo (Experimental): Participants received SoC daily PEX and SHP655 40 +/- 4 international units per kilogram (IU/kg), IV injection, QD, immediately after PEX and placebo 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
  Interventions: Other: Placebo; Drug: SHP655; Other: Standard of Care
- SoC + SHP655 (Experimental): Participants received SoC daily PEX and SHP655 40 +/- 4 IU/kg, IV injection, BID, immediately after PEX and 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
  Interventions: Drug: SHP655; Other: Standard of Care

INTERVENTIONS:
Other: Placebo — Participants will receive injection of placebo matched to SHP655.
  Arms: SoC + SHP655 + Placebo; Standard of Care (SoC) + Placebo
Drug: SHP655 — Participants will receive injection of SHP655.
  Other Names: rADAMTS-13
  Arms: SoC + SHP655; SoC + SHP655 + Placebo
Other: Standard of Care — Participants will receive PEX as Standard of Care (SOC).
  Other Names: PEX

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and efficacy of rADAMTS-13 (SHP655) administered in addition to standard of care (SoC) treatment of acquired thrombotic thrombocytopenic purpura (aTTP) participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant or legally authorized representative voluntarily signs informed consent. For participants unable to provide consent, a fully recognized medical proxy may be used according to local laws.
* Participant is 18 to 75 years old at the time of screening.
* Participant has been diagnosed with primary or secondary autoimmune acquired thrombotic thrombocytopenic purpura (aTTP) based on the following criteria:

  a) Thrombocytopenia [drop in platelet count >=50% or platelet count <100,000/microlitre (μL)] i) No more than 3 participants per arm may be enrolled with a screening platelet count >= 50,000/μL.

  b) Microangiopathic hemolytic anemia [elevation of lactate dehydrogenase (LDH) >2-fold or by presence or increase of schistocytes in peripheral blood smear].
* Willingness to fully comply with study procedures and requirements, and intention to initiate plasma exchange (PEX). Participants may be provisionally entered into the trial and undergo randomization pending the results of the ADAMTS-13 activity, anti-ADAMTS-13 antibody, and genetic testing for congenital thrombotic thrombocytopenic purpura (cTTP).
* If female of childbearing potential, participant presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study. Sexually active males must use an accepted and effective method of contraception during the treatment and until a minimum of 16 days after the last dose administered.

Exclusion Criteria:

* Participant has been diagnosed with congenital TTP.
* Participant has plasma ADAMTS-13 activity > 10% of normal at the central lab; if screening samples are not taken until after the first PEX, ADAMTS-13 activity from the local lab is permitted to determine eligibility.
* Participant has been diagnosed with another cause of thrombotic microangiopathy (TMA) including: DIC, disseminated malignancy, malignant hypertension, hematopoietic stem cell transplantation, shiga toxin related and atypical HUS, drug toxicity (e.g. gemcitabine, mitomycin C, clopidogrel) and pregnancy-related thrombocytopenia syndromes (e.g. HELLP, eclampsia).
* Participant has been exposed to another IP within 30 days prior to enrollment or is scheduled to participate in another clinical study involving IP or investigational device during the course of the study.
* Participant has received caplacizumab within 1 month prior to study enrollment.
* Participant is human immunodeficiency virus positive (HIV+) with unstable disease or CD4+ count <=200 cells/mm^3 within 3 months screening.
* Participants with conditions of severe immunodeficiency.
* Participant has had a previous aTTP event in the past 30 days.
* Participant has another underlying progressive fatal disease and/or life expectancy of less than 3 months.
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures
* Participant suffers from a mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude. However, a fully recognized medical proxy will be permitted to provide consent.
* If female, participant is pregnant or lactating.
* Participant is a family member or employee of the Sponsor or investigator.
* Any contraindication to PEX, methylprednisolone and/or rituximab as per prescribing information.
* Known life-threatening hypersensitivity reaction, including anaphylaxis, to the parent molecule ADAMTS-13, hamster protein, or other constituents of SHP655.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (24):
- United States (7):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
- Canada (2):
  - London Health Sciences Centre (LHSC) - University Hospital, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- France (4):
  - CHU de Reims - Hôpital Maison Blanche, Reims, Marne
  - Hopital Conception, Marseille
  - Chu Saint-Antoine, Paris
  - CHU de Rouen, Seine Maritime
- Hamatologie, Onkologie, Hämostaseologie, Frankfurt, Germany
- Italy (2):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Dr. Peset, Valencia
  - Hospital Universitari i Politècnic la Fe, Valencia
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, West Glamorgan
  - Royal Liverpool University Hospital, Liverpool
  - 1st Floor, UCLH-Haematology, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47aea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Canada, France, Great Britain, Spain and United States from 09 October 2019 to 05 August 2021.
Pre-assignment Details: Participants with a diagnosis of acquired thrombotic thrombocytopenic purpura (aTTP) were enrolled to receive placebo, SHP655 once daily (QD) and twice daily (BID) in a ratio of 1:1:1 in this study .
Groups:
- Standard of Care (SoC) + Placebo: Participants received SoC daily plasma exchange (PEX) followed by placebo immediately and 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
Period: Overall Study
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Started | 10 | 9 | 9
Pharmacokinetic Population (Pharmacokinetic (PK) set included all enrolled participants with confirmed aTTP diagnosis who have received at least 1 dose of investigational product and who have at least 1 evaluable post-dose PK value.) | 10 | 8 | 9
Completed | 9 | 6 | 8
Not Completed | 1 | 3 | 1
Not completed — Not Meeting Confirmatory Inclusion Criteria | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants randomized, who received any dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655 | Total
Number analyzed (Participants) | 10 | 9 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.80) | 51.9 (14.81) | 48.4 (14.93) | 47.0 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 5 | 19
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 8 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 1 | 0 | 1
  Race: Black or African American | 4 | 1 | 2 | 7
  Race: White | 6 | 5 | 6 | 17
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Other | 0 | 2 | 0 | 2
  Race: Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: ADAMTS-13 Activity Levels
Description: ADAMTS-13 Activity Levels was assessed by fluorescence resonance energy transfer (FRETS) ADAMTS13 activity, with or without SHP655 Supplementation. Schedule A (Days 1, 2, 3, 4, 6, 8, 11, and every 3 days thereafter) or Schedule B (Days 1, 2, 3, 5, 7, 9, 12, and every 3 days thereafter). Data is reported for multiple timepoints as Within 15 minutes pre-PEX and post-PEX; Within 15 minutes, 0.5-3 hours, 4-6 hours post end of investigational product (IP) infusion 1; Within 15 minutes, 0.5-3 hours post end IP infusion 2; 30 minutes pre-IP infusion 2 of Schedule A and Schedule B (up to Day 11 or 12).
Time Frame: Up to Days 11 or 12
Population: Pharmacokinetic (PK) Set included all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value (ADAMTS-13 antigen and ADAMTS-13 activity). Overall number analyzed are the number of participants available for analyses. Number analyzed are the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: international units(IU)/ml
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
international units(IU)/ml
  FRETS: Day 1: ≤15 min Pre-PEX: number analyzed (Participants) | 8 | 7 | 8
  FRETS: Day 1: ≤15 min Pre-PEX | 0.1439 (0.19247) | NA (NA) — Mean and Standard Deviation (SD) was not evaluable as the samples were below the lower limit of quantitation (LLOQ). | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 1: ≤15 min Post-PEX: number analyzed (Participants) | 9 | 8 | 9
  FRETS: Day 1: ≤15 min Post-PEX | 0.5418 (0.18345) | 0.5011 (0.19236) | 0.3029 (0.29020)
  FRETS: Day 1: ≤15 min Post End of IP 1: number analyzed (Participants) | 10 | 7 | 9
  FRETS: Day 1: ≤15 min Post End of IP 1 | 0.4571 (0.19125) | 2.012 (0.82832) | 1.352 (0.93502)
  FRETS: Day 1: 0.5-3 Hour (hr) Post End of IP 1: number analyzed (Participants) | 10 | 7 | 9
  FRETS: Day 1: 0.5-3 Hour (hr) Post End of IP 1 | 0.4420 (0.20895) | 1.905 (0.83349) | 1.266 (0.98904)
  FRETS: Day 1: 4-6 hr Post End of IP 1: number analyzed (Participants) | 10 | 5 | 9
  FRETS: Day 1: 4-6 hr Post End of IP 1 | 0.3197 (0.20545) | 1.163 (0.61343) | 0.7912 (0.69403)
  FRETS: Day 1: ≤30 min Pre-IP 2: number analyzed (Participants) | 10 | 6 | 9
  FRETS: Day 1: ≤30 min Pre-IP 2 | 0.2108 (0.19731) | 1.027 (0.55951) | 0.4949 (0.54891)
  FRETS: Day 1: ≤15 min Post End of IP 2: number analyzed (Participants) | 9 | 8 | 9
  FRETS: Day 1: ≤15 min Post End of IP 2 | 0.2267 (0.18660) | 1.022 (0.52060) | 1.545 (1.0854)
  FRETS: Day 1: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 8 | 7 | 9
  FRETS: Day 1: 0.5-3 hr Post End of IP 2 | 0.2007 (0.20012) | 1.015 (0.56462) | 1.300 (1.1114)
  FRETS: Day 2: ≤15 min Pre-PEX: number analyzed (Participants) | 10 | 7 | 8
  FRETS: Day 2: ≤15 min Pre-PEX | 0.1691 (0.15909) | 0.7650 (0.61929) | 0.9482 (0.99771)
  FRETS: Day 2: ≤15 min Post-PEX: number analyzed (Participants) | 10 | 7 | 9
  FRETS: Day 2: ≤15 min Post-PEX | 0.5801 (0.16107) | 0.7808 (0.36544) | 0.8426 (0.54317)
  FRETS: Day 2: ≤15 min Post End of IP 1: number analyzed (Participants) | 10 | 6 | 9
  FRETS: Day 2: ≤15 min Post End of IP 1 | 0.5433 (0.20267) | 1.965 (0.72122) | 1.977 (0.98427)
  FRETS: Day 2: 0.5-3 hr Post End of IP 1 | 0.5281 (0.24842) | 2.105 (1.0656) | 2.153 (1.3856)
  FRETS: Day 2: 4-6 hr Post End of IP 1: number analyzed (Participants) | 9 | 8 | 9
  FRETS: Day 2: 4-6 hr Post End of IP 1 | 0.4170 (0.25202) | 1.622 (0.78046) | 1.411 (0.75100)
  FRETS: Day 2: ≤30 min Pre-IP 2 | 0.3117 (0.24934) | 1.309 (0.48787) | 1.044 (0.55923)
  FRETS: Day 2: ≤15 min Post End of IP 2 | 0.2998 (0.24960) | 1.283 (0.52550) | 1.960 (0.99952)
  FRETS: Day 2: 0.5-3 hr Post End of IP 2 | 0.2833 (0.23999) | 1.398 (0.47591) | 2.129 (1.4547)
  FRETS: Day 3: ≤15 min Pre-PEX: number analyzed (Participants) | 9 | 6 | 5
  FRETS: Day 3: ≤15 min Pre-PEX | 0.2468 (0.23669) | 1.044 (0.54178) | 1.129 (1.0570)
  FRETS: Day 3: ≤15 min Post-PEX: number analyzed (Participants) | 10 | 8 | 6
  FRETS: Day 3: ≤15 min Post-PEX | 0.5342 (0.22251) | 0.7786 (0.16455) | 0.7020 (0.40432)
  FRETS: Day 3: ≤15 min Post End of IP 1: number analyzed (Participants) | 10 | 8 | 6
  FRETS: Day 3: ≤15 min Post End of IP 1 | 0.5215 (0.23522) | 2.210 (0.96057) | 1.911 (1.6633)
  FRETS: Day 3: 0.5-3 hr Post End of IP 1: number analyzed (Participants) | 10 | 8 | 6
  FRETS: Day 3: 0.5-3 hr Post End of IP 1 | 0.4970 (0.23979) | 2.086 (0.85567) | 1.785 (1.1566)
  FRETS: Day 3: 4-6 hr Post End of IP 1: number analyzed (Participants) | 10 | 8 | 7
  FRETS: Day 3: 4-6 hr Post End of IP 1 | 0.4670 (0.30646) | 1.680 (0.46457) | 1.271 (0.71567)
  FRETS: Day 3: ≤30 min Pre-IP 2: number analyzed (Participants) | 10 | 7 | 7
  FRETS: Day 3: ≤30 min Pre-IP 2 | 0.3424 (0.29275) | 1.196 (0.44550) | 1.041 (0.84152)
  FRETS: Day 3: ≤15 min Post End of IP 2: number analyzed (Participants) | 10 | 7 | 6
  FRETS: Day 3: ≤15 min Post End of IP 2 | 0.3514 (0.31264) | 1.263 (0.38468) | 1.478 (1.0343)
  FRETS: Day 3: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 10 | 7 | 7
  FRETS: Day 3: 0.5-3 hr Post End of IP 2 | 0.3227 (0.28191) | 1.267 (0.43580) | 1.902 (1.4522)
  FRETS: Day 4 or 5: ≤15 min Pre-PEX: number analyzed (Participants) | 7 | 6 | 5
  FRETS: Day 4 or 5: ≤15 min Pre-PEX | 0.2378 (0.30513) | 1.094 (0.67793) | 1.378 (1.1964)
  FRETS: Day 4 or 5: ≤15 min Post-PEX: number analyzed (Participants) | 7 | 8 | 5
  FRETS: Day 4 or 5: ≤15 min Post-PEX | 0.4554 (0.26405) | 0.8222 (0.21072) | 0.8725 (0.57834)
  FRETS: Day 4 or 5: ≤15 min Post End of IP 1: number analyzed (Participants) | 7 | 8 | 5
  FRETS: Day 4 or 5: ≤15 min Post End of IP 1 | 0.7599 (1.0062) | 2.257 (0.95791) | 1.679 (1.3803)
  FRETS: Day 4 or 5: 0.5-3 hr Post End of IP 1: number analyzed (Participants) | 7 | 8 | 5
  FRETS: Day 4 or 5: 0.5-3 hr Post End of IP 1 | 0.6699 (0.76875) | 2.425 (1.4869) | 1.405 (1.0118)
  FRETS: Day 4 or 5: 4-6 hr Post End of IP 1: number analyzed (Participants) | 7 | 7 | 5
  FRETS: Day 4 or 5: 4-6 hr Post End of IP 1 | 0.5663 (0.69581) | 1.741 (0.84171) | 1.214 (1.0280)
  FRETS: Day 4 or 5: ≤30 min Pre-IP 2: number analyzed (Participants) | 6 | 6 | 5
  FRETS: Day 4 or 5: ≤30 min Pre-IP 2 | 0.5045 (0.60730) | 1.290 (0.64745) | 1.255 (0.98796)
  FRETS: Day 4 or 5: ≤15 min Post End of IP 2: number analyzed (Participants) | 6 | 6 | 5
  FRETS: Day 4 or 5: ≤15 min Post End of IP 2 | 0.4596 (0.58498) | 1.288 (0.63801) | 2.306 (1.6006)
  FRETS: Day 4 or 5: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 6 | 6 | 5
  FRETS: Day 4 or 5: 0.5-3 hr Post End of IP 2 | 0.4129 (0.49574) | 1.106 (0.59034) | 2.009 (1.4354)
  FRETS: Day 6 or 7: ≤15 min Pre-PEX: number analyzed (Participants) | 4 | 2 | 2
  FRETS: Day 6 or 7: ≤15 min Pre-PEX | 0.1246 (0.24910) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: ≤15 min Post-PEX: number analyzed (Participants) | 4 | 3 | 2
  FRETS: Day 6 or 7: ≤15 min Post-PEX | 0.2587 (0.30131) | 0.7311 (0.48855) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: ≤15 min Post End of IP 1: number analyzed (Participants) | 4 | 3 | 2
  FRETS: Day 6 or 7: ≤15 min Post End of IP 1 | 0.2150 (0.26924) | 1.481 (0.89773) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: 0.5-3 hr Post End of IP 1: number analyzed (Participants) | 4 | 3 | 2
  FRETS: Day 6 or 7: 0.5-3 hr Post End of IP 1 | 0.2194 (0.24929) | 1.673 (1.0721) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: 4-6 hr Post End of IP 1: number analyzed (Participants) | 4 | 3 | 2
  FRETS: Day 6 or 7: 4-6 hr Post End of IP 1 | 0.1443 (0.24485) | 1.467 (1.1232) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: ≤30 min Pre-IP 2: number analyzed (Participants) | 4 | 2 | 2
  FRETS: Day 6 or 7: ≤30 min Pre-IP 2 | 0.1272 (0.25440) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: ≤15 Minutes Post End of IP 2: number analyzed (Participants) | 4 | 2 | 2
  FRETS: Day 6 or 7: ≤15 Minutes Post End of IP 2 | 0.1422 (0.28435) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  FRETS: Day 6 or 7: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 4 | 2 | 1
  FRETS: Day 6 or 7: 0.5-3 hr Post End of IP 2 | 0.1336 (0.26710) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not estimable for 1 participant.
  FRETS: Day 8 or 9: ≤15 min Pre-PEX: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: ≤15 min Pre-PEX |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: ≤15 min Post-PEX: number analyzed (Participants) | 0 | 2 | 0
  FRETS: Day 8 or 9: ≤15 min Post-PEX |  | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. |
  FRETS: Day 8 or 9: ≤15 min Post End of IP 1: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: ≤15 min Post End of IP 1 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: 0.5-3 hr Post End of IP 1: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: 0.5-3 hr Post End of IP 1 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: 4-6 hr Post End of IP 1: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: 4-6 hr Post End of IP 1 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: ≤30 Minutes Pre-IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: ≤30 Minutes Pre-IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: ≤15 min Post End of IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: ≤15 min Post End of IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 8 or 9: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9: 0.5-3 hr Post End of IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: ≤15 min Pre-PEX: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 11 or 12: ≤15 min Pre-PEX |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: ≤15 min Post-PEX: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 11 or 12: ≤15 min Post-PEX |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: ≤15 min Post End of IP 1: number analyzed (Participants) | 0 | 0 | 0
  FRETS: Day 11 or 12: 0.5-3 hr Post End of IP 1: number analyzed (Participants) | 0 | 0 | 0
  FRETS: Day 11 or 12: 4-6 hr Post End of IP 1: number analyzed (Participants) | 0 | 0 | 0
  FRETS: Day 11 or 12: ≤30 min Pre-IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 11 or 12: ≤30 min Pre-IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: ≤15 min Post End of IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 11 or 12: ≤15 min Post End of IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: 0.5-3 hr Post End of IP 2: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 11 or 12: 0.5-3 hr Post End of IP 2 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |

2. Primary Outcome: Platelet Count
Description: The platelet counts are reported in units of 10^9 per liter blood.
Time Frame: Baseline and end of study (EOS) (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product. Overall number analyzed are the number of participants with data evaluable for analyses. Number analyzed is the number of participants available for analysis.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Groups:
- SoC + SHP655 + Placebo: Participants received SoC daily PEX and SHP655 40 +/- 4 IU/kg, IV injection, QD, immediately after PEX and placebo 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
10^9 platelets/L
  Baseline | 35.80 (32.076) | 27.67 (17.571) | 15.38 (7.463)
  EOS: number analyzed (Participants) | 9 | 7 | 9
  EOS | 278.89 (79.592) | 267.00 (86.906) | 286.22 (109.264)

3. Primary Outcome: Lactate Dehydrogenase (LDH) Levels
Description: The lactate dehydrogenase levels are reported.
Time Frame: Baseline and EOS (up to approximately 15 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: international units (IU)/L
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 8
international units (IU)/L
  Baseline | 634.6 (378.37) | 616.3 (478.14) | 787.8 (188.39)
  EOS: number analyzed (Participants) | 8 | 6 | 8
  EOS | 197.3 (42.00) | 208.8 (75.20) | 220.4 (69.93)

4. Secondary Outcome: Dose(s) of SHP655 Needed to Achieve and Maintain Adequate Plasma Levels of rADAMTS-13
Description: Dose(s) of SHP655 needed to achieve and maintain adequate plasma levels of rADAMTS-13 in order to support induction of remission and to reduce the number of PEX procedures needed for the treatment of acute aTTP episodes was assessed.
Time Frame: From start of study drug administration up to 13 weeks (following remission up to 6 months)
Population: Data could not be analyzed due to sparse sample collections and confounding dosing inputs with daily sequential PEX + SHP655 dosing.
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: PK/PD Temporal Relationship of Safety and Efficacy Parameter as a Function of ADAMTS-13 Activity
Description: Parameters included platelet and LDH counts.
Time Frame: Up to 6 months
Population: as for outcome 4
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With ADAMTS-13 Binding Antibodies Per Titer
Description: Antibody titer indicates the level of the antibodies in a blood sample, defined as the greatest dilution (or lowest concentration) of the blood sample at which an antibody assay (such as ELISA for e.g.), still produces a detectable positive result. Data is presented per titer for ADA positive participants only.
Time Frame: Baseline and EOS (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product. Overall number analyzed are the number of participants are ADA positive participants. Number analyzed is the number of participants available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- SoC + SHP655 + Placebo: Participants received SoC daily PEX and SHP655 40 +/- 4 international IU/kg, IV injection, QD, immediately after PEX and placebo 12 +/- 1 hours after completion of PEX until remission was achieved (up to approximately 6 months).
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 7 | 8 | 8
Participants
  Baseline- 1:20 | 2 | 3 | 1
  Baseline- 1:40 | 3 | 2 | 2
  Baseline- 1:80 | 2 | 0 | 1
  Baseline- 1:160 | 0 | 1 | 2
  Baseline- 1:320 | 0 | 2 | 0
  Baseline- 1:640 | 0 | 0 | 1
  Baseline- 1:1280 | 0 | 0 | 1
  EOS- 1:20: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:20 | 0 | 1 | 0
  EOS- 1:40: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:40 | 2 | 0 | 1
  EOS- 1:80: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:80 | 1 | 0 | 2
  EOS- 1:2560: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:2560 | 0 | 1 | 0
  EOS- 1:5120: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:5120 | 0 | 0 | 1
  EOS- 1:81920: number analyzed (Participants) | 3 | 2 | 5
  EOS- 1:81920 | 0 | 0 | 1

7. Secondary Outcome: Inhibitory Autoantibodies (Nab) Titer Levels
Description: NAb titers were summarized (median, minimum and maximum) at baseline and EOS per treatment arms, in those subjects with NAb positive results (NAb positive is defined as titer value >=0.6 BU/mL).
Time Frame: Baseline and EOS (up to approximately 15 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: BU/mL
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
BU/mL
  Baseline | 1.25 [0.6 to 3.4] | 1.25 [1.0 to 1.8] | 1.80 [0.6 to 4.0]
  EOS: number analyzed (Participants) | 9 | 7 | 8
  EOS | 0.60 [0.6 to 0.6] | 0.70 [0.7 to 1.7] | 4.00 [4.0 to 4.0]

8. Secondary Outcome: ADAMTS-13 Activity Levels in Participants Receiving Additional SHP655 for up to 30 Days After Resolution by Using FRETS
Description: ADAMTS-13 activity levels in participants receiving additional SHP655 for up to 30 days after the resolution of the thrombotic thrombocytopenic purpura (TTP) episode were assessed. Resolution was defined as a normal platelet count and LDH <2 ULN for at least 48 hours following initial normalization of platelet count (acute episode period).
Time Frame: At Days 3, 7, 10, 21, 28, 42, 56 and 84
Population: PK Set included all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value (ADAMTS-13 antigen and ADAMTS-13 activity). Overall number analyzed are the number of participants available for analyses. Number analyzed is the number of participants with data available for analyses at given time point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 7 | 7 | 6
IU/mL
  Day 3: number analyzed (Participants) | 6 | 2 | 6
  Day 3 | 0.4602 (0.14328) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | 0.1171 (0.28688)
  Day 7: number analyzed (Participants) | 4 | 7 | 2
  Day 7 | 0.3037 (0.26921) | 0.3180 (0.34714) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  Day 10: number analyzed (Participants) | 3 | 4 | 5
  Day 10 | 0.9021 (0.20520) | 0.5518 (0.33962) | 0.4904 (0.46441)
  Day 21: number analyzed (Participants) | 4 | 5 | 5
  Day 21 | 0.8102 (0.52773) | 0.6264 (0.60971) | 0.5320 (0.51432)
  Day 28: number analyzed (Participants) | 4 | 5 | 4
  Day 28 | 0.8830 (0.51516) | 0.8931 (0.41323) | 0.8632 (0.62848)
  Day 42: number analyzed (Participants) | 4 | 4 | 4
  Day 42 | 0.9968 (0.36745) | 0.8842 (0.39784) | 1.055 (0.36080)
  Day 56: number analyzed (Participants) | 3 | 4 | 3
  Day 56 | 1.088 (0.25524) | 0.9923 (0.33663) | 1.092 (0.19961)
  Day 84: number analyzed (Participants) | 7 | 6 | 6
  Day 84 | 0.9708 (0.43831) | 1.021 (0.65715) | 0.6051 (0.48113)

9. Secondary Outcome: Relationship Between ADAMTS-13 Activity and End-organ Disease Status
Description: End-organ disease status were evaluated for renal, cardiac and neurological diseases.
Time Frame: Up to 6 months
Population: as for outcome 4
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Predose Concentration (Cpre) to Maximum Plasma Concentration (Cmax) Ratio
Time Frame: Pre-PEX and post-PEX at multiple timepoints at Days 1, 2, 3, 4 or 5, 6 or 7, 8 or 9, and 11 or 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 7 | 7 | 9
ratio
  FRETS: Day 1: number analyzed (Participants) | 5 | 2 | 1
  FRETS: Day 1 | 2.744 (3.3837) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not estimable for 1 participant.
  FRETS: Day 2: number analyzed (Participants) | 4 | 7 | 7
  FRETS: Day 2 | 2.587 (0.92176) | 3.534 (2.4373) | 3.675 (2.3380)
  FRETS: Day 3: number analyzed (Participants) | 4 | 7 | 6
  FRETS: Day 3 | 1.669 (0.34045) | 2.134 (0.45392) | 2.268 (1.0679)
  FRETS: Day 4 or 5: number analyzed (Participants) | 2 | 5 | 5
  FRETS: Day 4 or 5 | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | 2.543 (0.59576) | 1.972 (0.91248)
  FRETS: Day 6 or 7: number analyzed (Participants) | 1 | 2 | 1
  FRETS: Day 6 or 7 | NA (NA) — Mean and SD was not estimable for 1 participant. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not estimable for 1 participant.
  FRETS: Day 8 or 9: number analyzed (Participants) | 0 | 1 | 0
  FRETS: Day 8 or 9 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  FRETS: Day 11 or 12: number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: AUC Overall: Area Under the Plasma Concentration Time Curve ADAMTS13 Activity by Using FRETS
Time Frame: Within 15 min pre-PEX and at multiple timepoints Post PEX at Days 1, 2, 3, 4 or 5 and 6 or 7
Population: PK Set included all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value (ADAMTS-13 antigen and ADAMTS-13 activity). Number analyzed are the number of participants available for analysis at the specific time point.
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
h*IU/mL
  Day 1: number analyzed (Participants) | 9 | 7 | 8
  Day 1 | 3.563 (2.5551) | 19.87 (9.1150) | 12.80 (8.4633)
  Day 2 | 4.461 (3.9480) | 24.16 (9.0323) | 21.97 (11.135)
  Day 3: number analyzed (Participants) | 9 | 7 | 6
  Day 3 | 5.590 (4.7232) | 22.75 (5.6549) | 23.49 (9.2589)
  Day 4 or 5: number analyzed (Participants) | 5 | 6 | 5
  Day 4 or 5 | 9.507 (11.592) | 24.10 (11.357) | 22.05 (14.192)
  Day 6 or 7: number analyzed (Participants) | 2 | 2 | 2
  Day 6 or 7 | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ. | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.

12. Secondary Outcome: Systemic and Antibody Induced Clearance
Time Frame: 15 minutes pre-PEX,15 minutes post-PEX,15 minutes, 0.5-3 hours, 4-6 hours post end of IP infusion 1,30 minutes pre-IP infusion 2,15 minutes, 0.5-3 hours post-IP infusion 2 of Schedule A or Schedule B (up to 6 months)
Population: as for outcome 4
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Cmax: Maximum ADAMTS-13 Activity Between PEX or SHP655 Infusions by Using FRETS
Time Frame: Pre-PEX and post-PEX at multiple timepoints at Days 1, 2, 3, 4 or 5, 6 or 7, 8 or 9, and 11 or 12
Population: PK Set included all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value (ADAMTS-13 antigen and ADAMTS-13 activity). Number analyzed is the number of participants available for analyses at given time point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
IU/mL
  Day 1: number analyzed (Participants) | 10 | 7 | 9
  Day 1 | 0.4157 (0.17075) | 2.011 (0.79036) | 1.653 (1.0655)
  Day 2: number analyzed (Participants) | 10 | 7 | 9
  Day 2 | 0.4951 (0.27178) | 2.153 (1.1404) | 2.458 (1.4369)
  Day 3: number analyzed (Participants) | 10 | 8 | 7
  Day 3 | 0.4307 (0.28420) | 2.228 (0.93968) | 2.222 (1.5080)
  Day 4 or 5: number analyzed (Participants) | 7 | 7 | 5
  Day 4 or 5 | 0.6438 (0.97767) | 2.633 (1.4955) | 2.377 (1.5934)
  Day 6 or 7: number analyzed (Participants) | 4 | 3 | 2
  Day 6 or 7 | 0.1362 (0.095283) | 1.625 (1.0126) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.
  Day 8 or 9: number analyzed (Participants) | 0 | 1 | 0
  Day 8 or 9 |  | NA (NA) — Mean and SD was not estimable for 1 participant. |
  Day 11 or 12: number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Trough Levels of ADAMTS-13 Prior PEX ADAMTS13 Activity by Using FRETS
Time Frame: Within 15 min pre-PEX and at multiple timepoints Post PEX at Days 2, 3, 4 or 5 and 6 or 7
Population: PK Set included all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value (ADAMTS-13 antigen and ADAMTS-13 activity). Overall number analyzed are the number of participants available for analyses. Number analyzed are the number of participants with data available for analysis at the specific time point.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 7 | 8 | 9
IU/mL
  Day 2 | 0.1667 (0.17308) | 0.8493 (0.62139) | 0.9274 (0.93426)
  Day 3: number analyzed (Participants) | 7 | 7 | 7
  Day 3 | 0.2579 (0.26836) | 1.110 (0.52612) | 1.174 (0.93910)
  Day 4 or 5: number analyzed (Participants) | 4 | 7 | 5
  Day 4 or 5 | 0.3138 (0.38416) | 1.180 (0.65905) | 1.378 (1.1976)
  Day 6 or 7: number analyzed (Participants) | 3 | 3 | 2
  Day 6 or 7 | 0.1660 (0.28752) | 1.070 (0.98879) | NA (NA) — Mean and SD was not evaluable as the samples were below LLOQ.

15. Secondary Outcome: Percentage of Participants With ADAMTS-13 Activity Trough Levels >10%
Time Frame: Pre-dose at Days 2, 3 4 or 5, 6 or 7, 8 or 9, and 11 or 12
Population: PK Set:all enrolled participants with confirmed aTTP diagnosis who received at least 1 dose of investigational product and who had at least 1 evaluable post-dose PK value.Overall number:particiapnts from PK set,included number of participants available for analysis.Number analyzed:number of participants available with ADAMTS activity absolute Ctrough values at given time point.Percentages are calculated based on total number of participants available for corresponding stratification per day.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 7 | 8 | 9
percentage of participants
  Day 2 | 57.1 | 100.0 | 77.8
  Day 3: number analyzed (Participants) | 7 | 7 | 7
  Day 3 | 57.1 | 100.0 | 85.7
  Day 4 or 5: number analyzed (Participants) | 4 | 6 | 5
  Day 4 or 5 | 50.0 | 100.0 | 100.0
  Day 6 or 7: number analyzed (Participants) | 3 | 3 | 2
  Day 6 or 7 | 33.3 | 66.7 | 50.0
  Day 8 or 9: number analyzed (Participants) | 0 | 1 | 0
  Day 8 or 9 |  | 100.0 |
  Day 11 or 12: number analyzed (Participants) | 0 | 1 | 0
  Day 11 or 12 |  | 100.0 |

16. Secondary Outcome: Number of Participants Who Achieved Remission Following Normalization of Platelet Count
Description: Remission was defined as the time taken to achieve platelet count ≥150,000/μL, which was confirmed by a second normal platelet count ≥150,000/μL and LDH <2 ULN 48 hours following initial normalization.
Time Frame: From the start of study drug administration up to 6 months post remission
Population: FAS included all enrolled participants with confirmed aTTP diagnosis who were treated with a study product and had an ADAMTS-13 activity reading from at least one post infusion sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
Participants | 9 | 8 | 8

17. Secondary Outcome: Percentage of Participants Achieving Remission
Description: Remission was defined as a normal platelet count and LDH <2 upper limit of normal (ULN) for at least 48 hours following initial normalization of platelet count (acute episode period). Normalization of platelet count was defined ≥150,000/μL, which was confirmed by a second normal platelet count ≥150,000/μL and LDH <2 ULN.
Time Frame: From the start of study drug administration up to 6 months post remission
Population: FAS included all enrolled participants with confirmed aTTP diagnosis who were treated with a study product and had an ADAMTS-13 activity reading from at least one post infusion sample. Overall number analyzed are the number of participants with data evaluable for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 8
percentage of participants | 100.0 [69.15 to 100.00] | 100.0 [63.06 to 100.00] | 88.9 [51.75 to 99.72]

18. Secondary Outcome: Time to First Exacerbation
Description: Exacerbation was defined as recurrent thrombocytopenia following a response and requiring a reinitiation of daily plasma exchange treatment after ≥1 day but ≤30 days of no plasma exchange treatment. Data is reported based on Kaplan-Meier estimates. Data was reported for time to first exacerbation in categories for participants enrolled before protocol amendment 4 (from study start up to 11 months) and after protocol amendment 4 (from 11 months up to the EOS).
Time Frame: From start of study drug administration up to EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Median (50% Confidence Interval); unit: days
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
days
  From Study Start up to 11 Months | NA [2.00 to NA] — The median and upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | 8.0 [5.00 to NA] — The upper limit of CI was not estimable due to insufficient number of participants with events.
  From 11 Months up to EOS (up to approximately 15 months) | NA [4.00 to NA] — The median and upper limit of CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | NA [6.00 to NA] — The median and upper limit of CI was not estimable due to insufficient number of participants with events.

19. Secondary Outcome: Time to Relapse
Description: Relapse was determined by platelet count or the occurrence after remission of a major clinical event (e.g., Myocardial Infraction (MI), stroke, death) deemed by the investigator to be related to aTTP. Data was reported for time to relapse in categories for participants enrolled before protocol amendment 4 (from study start up to 11 months) and after protocol amendment 4 (from 11 months up to the EOS).
Time Frame: From start of study drug administration up to EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Median (50% Confidence Interval); unit: days
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
days
  From Study Start up to 11 Months | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants.
  From 11 Months up to EOS (up to approximately 15 months) | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants. | NA [NA to NA] — The median, lower and upper limit of CI was not evaluable due to no events in participants.

20. Secondary Outcome: Percentage of Participants With Exacerbation
Description: Exacerbation was determined by platelet count or the occurrence after remission of a major clinical event (e.g., myocardial infarction (MI), stroke, death) deemed by the investigator to be related to aTTP. Data was reported for percentage of participants with exacerbation in categories for participants enrolled before protocol amendment 4 (from study start up to 11 months) and after protocol amendment 4 (from 11 months up to the EOS).
Time Frame: From start of study drug administration up to EOS (up to approximately 15 months)
Population: FAS included all enrolled participants with confirmed aTTP diagnosis who were treated with a study product and had an ADAMTS-13 activity reading from at least one post infusion sample. Overall number of participants analyzed are number of participants achieving remission. Number analyzed are the number of participants with data available for analyses at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 8
percentage of participants
  From Study Start up to 11 Months: number analyzed (Participants) | 4 | 4 | 5
  From Study Start up to 11 Months | 50.0 [6.76 to 93.24] | 0.0 [0.00 to 60.24] | 60.0 [14.66 to 94.73]
  From 11 Months up to EOS (up to approximately 15 months): number analyzed (Participants) | 6 | 4 | 3
  From 11 Months up to EOS (up to approximately 15 months) | 33.3 [4.33 to 77.72] | 0.0 [0.00 to 60.24] | 33.3 [0.84 to 90.57]

21. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was determined by platelet count or the occurrence after remission of a major clinical event (e.g., Myocardial Infraction (MI), stroke, death) deemed by the investigator to be related to aTTP. Data was reported for percentage of participants with exacerbation in categories for participants enrolled before protocol amendment 4 (from study start up to 11 months) and after protocol amendment 4 (from 11 months up to the EOS).
Time Frame: From start of study drug administration up to EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
percentage of participants
  From Study Start up to 11 Months | 0.0 [0.0 to 60.24] | 0.0 [0.0 to 60.24] | 0.0 [0.0 to 52.18]
  From 11 Months up to EOS (up to approximately 15 months) | 0.0 [0.0 to 45.93] | 0.0 [0.0 to 60.24] | 0.0 [0.0 to 70.76]

22. Secondary Outcome: Percentage of Participants With Major Clinical Events Related to Thrombotic Thrombocytopenic Purpura (TTP)
Description: Major clinical events related to TTP included Death, Stroke, MI and organ dysfunction not normalized within the 90-day observation period which consisted of chronic renal insufficiency, neurologic impairment and neurocognitive deficits.
Time Frame: From start of study drug administration up to EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
percentage of participants
  Renal Insufficiency | 90.0 | 100.0 | 88.9
  Neurologic Deficits | 60.0 | 100.0 | 77.8
  Brain Injury | 50.0 | 62.5 | 66.7
  Death, Stroke and MI | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Major Clinical Events Related to PEX
Description: Major clinical events included clinically relevant bleeding (modified ITP score) or thrombosis at the site of line insertion, adverse reactions to plasma, including citrate reactions, allergic reactions, and transfusion-related acute lung injury (TRALI). Data is reported by summarizing the data for all parameters.
Time Frame: Up to 6 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
Participants | 6 | 1 | 1

24. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Titer of Binding Relative to Baseline
Time Frame: Baseline and EOS (at approximately Month 15)
Population: SAS included all participants randomized, who received any dose of investigational product. Overall number analyzed are the number of participants available for analyses. Number analyzed are the number of participants with data available for analysis at the specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants
  Baseline | 7 | 8 | 8
  EOS at Month 15: number analyzed (Participants) | 9 | 7 | 8
  EOS at Month 15 | 3 | 2 | 5

25. Secondary Outcome: Number of Participants With Inhibitory Antibodies Relative to Baseline
Time Frame: Baseline and EOS (at approximately Month 15)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants
  Baseline | 6 [0.6 to 3.4] | 4 [1.0 to 1.8] | 7 [0.6 to 4.0]
  EOS at Month 15: number analyzed (Participants) | 9 | 7 | 8
  EOS at Month 15 | 3 [0.6 to 0.6] | 3 [0.7 to 1.7] | 2 [4.0 to 4.0]

26. Secondary Outcome: Percentage of Participants With at Least One Positive Identification of Antibodies to SHP655
Description: Percentages are based on the total number of participants per treatment group that have at least one ADA sample analyzed.
Time Frame: Up to 6 months
Population: Full Analysis Set (FAS) included all enrolled participants with confirmed aTTP diagnosis who were treated with a study product and had an ADAMTS-13 activity reading from at least one post infusion sample.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
percentage of participants
  ADA Positive: up to 3 Months | 80.0 | 62.5 | 88.9
  ADA Positive: up to 6 Months | 20.0 | 75.0 | 33.3
  Nab Positive: up to 3 Months | 40.0 | 37.5 | 33.3
  Nab Positive: up to 6 Months | 30.0 | 37.5 | 22.2

27. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Specifically Product-Related TEAEs and Serious TEAEs
Description: AE=any untoward medical occurrence in a participants administered IP that does not necessarily have a causal relationship with the treatment. TEAE=an adverse event with an onset that occurs after receiving study drug. SAE=an AE with any untoward clinical manifestation of signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, important medical event, bronchospasm associated with anaphylaxis, reviewed and confirmed seroconversion for human immunodeficiency virus (HIV), hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), hepatitis E virus (HEV), or parvovirus B19 (B19V). A product related AE is any event emerging or manifesting at or after the initiation of treatment with an investigational product or medicinal product or any existing event that worsens.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants
  Any TEAEs | 10 | 9 | 8
  Specifically Product-Related TEAEs | 0 | 1 | 0
  Serious TEAEs | 4 | 1 | 3

28. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Vital Signs
Description: Vital signs were assessed based on blood pressure, pulse rate, respiratory rate and body temperature.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Clinical Chemistry
Description: Clinical chemistry assessed alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase, blood urea nitrogen, creatinine, and glucose.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Hematology
Description: Hematology consisted of complete blood count and leukocytes with differential (basophils, eosinophils, lymphocytes, monocytes, neutrophils), mean corpuscular volume (MCV), mean corpuscular hemoglobin concentration (MCHC) and platelet count.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: SAS included all participants randomized, who received any dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 9 | 9
Participants | 0 | 0 | 0

31. Secondary Outcome: Percentage of Participants Receiving Rescue Therapy
Description: Rescue therapy was defined as any product with a known interruption to the pharmacokinetic/ pharmacodynamic (PK/PD) relationship between ADAMTS-13 activity, von Willebrand factor (VWF) activity, and platelet count. If rescue therapy was initiated, the administration of IP (SHP655 or placebo) was suspended for the duration of the study. Number of participants experiencing occurrence of receiving rescue therapy was assessed.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
percentage of participants | 20.0 | 0 | 22.2

32. Secondary Outcome: Percentage of Participants Meeting Rescue Criteria
Description: Rescue therapy was defined as any product with a known interruption to the PK/PD relationship between ADAMTS-13 activity, VWF activity, and platelet count. If rescue therapy was initiated, the administration of IP (SHP655 or placebo) was suspended for the duration of the study. Number of participants experiencing occurrence in meeting rescue therapy criteria was assessed. Percentage of participants with rescue therapy initiated are based on laboratory criteria and adverse events.
Time Frame: From first dose of study drug until the EOS (up to approximately 15 months)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) + Placebo | SoC + SHP655 + Placebo | SoC + SHP655
Number analyzed (Participants) | 10 | 8 | 9
percentage of participants | 10.0 | 0.0 | 11.1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of the study (up to approximately 15 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Placebo Post PEX + Placebo 12H Post PEX: Placebo Post PEX + Placebo 12H Post PEX
- SHP655 40 IU/kg Post PEX + Placebo 12H Post PEX: SHP655 40 IU/kg Post PEX + Placebo 12H Post PEX
- SHP655 40 IU/kg Post PEX + SHP655 40 IU/kg 12H Post PEX: SHP655 40 IU/kg Post PEX + SHP655 40 IU/kg 12H Post PEX
Arm/Group | Placebo Post PEX + Placebo 12H Post PEX | SHP655 40 IU/kg Post PEX + Placebo 12H Post PEX | SHP655 40 IU/kg Post PEX + SHP655 40 IU/kg 12H Post PEX
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/9 | 3/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Post PEX + Placebo 12H Post PEX (N=10) | SHP655 40 IU/kg Post PEX + Placebo 12H Post PEX (N=9) | SHP655 40 IU/kg Post PEX + SHP655 40 IU/kg 12H Post PEX (N=9)
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Post PEX + Placebo 12H Post PEX (N=10) | SHP655 40 IU/kg Post PEX + Placebo 12H Post PEX (N=9) | SHP655 40 IU/kg Post PEX + SHP655 40 IU/kg 12H Post PEX (N=9)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1
Anal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 1
Catheter site pain (General disorders) | 2 | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0
Citrate toxicity (Injury, poisoning and procedural complications) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 1
Heart rate increased (Investigations) | 0 | 2 | 0
Hot flush (Vascular disorders) | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Medical device site discomfort (General disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1 | 0
Peripheral swelling (General disorders) | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Procedural anxiety (Psychiatric disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Pyrexia (General disorders) | 3 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin weeping (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Swelling face (General disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Transfusion related complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
White blood cell count abnormal (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (6):
  • Study Protocol: Original (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/Prot_000.pdf
  • Study Protocol: Protocol Amendment 1 (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/Prot_001.pdf
  • Study Protocol: Protocol Amendment 2 (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/Prot_002.pdf
  • Study Protocol: Protocol Amendment 3 (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/Prot_003.pdf
  • Study Protocol: Protocol Amendment 4 (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/Prot_004.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03922308/SAP_005.pdf